CLINICAL TRIAL: NCT01245257
Title: Effects of Prednisolone and Pentoxifylline on the Regulation of Urea Synthesis in Alcoholic Hepatitis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: FHNC-Alk-Hep
Record Dates: First submitted 2010-11-15; First posted 2010-11-22 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2013-12

CONDITIONS: Alcoholic Hepatitis
Keywords: Inflammation; Urea Synthesis; Catabolism; Nitrogen balance
MeSH Terms: conditions — Hepatitis, Alcoholic; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alcoholic Hepatitis: Patients with alcoholic hepatitis

SUMMARY:
Loss of total mass of muscles (catabolism) is a serious clinical problem in patients with alcoholic hepatitis. The liver might play an important role in this stress-catabolism by increasing the production of urea during the inflammatory process.

The purpose of this study is to examine the regulation of urea synthesis in patients with alcoholic hepatitis and to study the effect of the anti-inflammatory drugs prednisolone and pentoxifylline on this regulation.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic hepatitis (alcohol intake (> 40g/day in 6 months), bilirubin > 80 μmol/l)

Exclusion Criteria:

* Severe bacterial infections
* Other chronical inflammatory diseases
* Cancer
* Other catabolic diseases
* Treatment with prednisolone or pentoxifylline within the last 8 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with alcoholic hepatitis admitted to hospital for treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Functional Hepatic Nitrogen Clearance | At inclusion, after approximately 3 month and if severe alcoholic hepatitis also after 14 days medical treatment

SECONDARY OUTCOMES:
Clinical and biochemical measures of inflammation | At inclusion, after approximately 3 month and if severe alcoholic hepatitis also after 14 days medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen Louise Thomsen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Medicine V, Aarhus University Hospital, Aarhus, Denmark